CLINICAL TRIAL: NCT01980719
Title: Molecular Determinants of Persistent Cancer Related Fatigue
Acronym: MDOF
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Suzanna Zick, Research Associate Professor, University of Michigan
Other Study IDs: HUM00038766
Record Dates: First submitted 2013-10-29; First posted 2013-11-11 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2013-11

CONDITIONS: Fatigue; Pain; Poor Sleep Quality
MeSH Terms: conditions — Fatigue; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy, Age-Matched
- Fatigued
- Not Fatigued

SUMMARY:
The purpose of this study is to determine if inflammatory markers in blood as well as brain neurotransmitters (markers of in-brain activity and metabolism) are related to long-term or chronic fatigue.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

- Women age 18 or older with no contraindication to magnetic resonance imaging(MRI);

Fatigued BC Participants:

* Have a diagnosis of breast cancer;
* And have completed all cancer-related treatments (i.e., surgery, chemotherapy, radiotherapy, immunotherapy, etc.) except for hormonal therapy and or herceptin at least 12 weeks previously; and be apparently cancer-free.

Age-Matched, Healthy Participants:

* Generally healthy;
* Matched in age ± 2.5 years to a Fatigued BC participant.
* No prior history of any cancer except for basal cell or squamous cell tumors of the skin that have been surgically excised;
* Have good sleep quality
* Have no chronic pain
* Have no chronic fatigue

Exclusion Criteria:

* Pregnant, wanting to become pregnant or lactating women ;
* Diagnosed with anemia [defined as hemoglobin levels < 12 gm/dl] or receiving treatment for anemia ;
* Diagnosed with any comorbidities likely to cause significant fatigue (i.e., moderate to severe heart failure)
* Diagnosed with nutritional deficiencies;
* Have a diagnosis of untreated hypo- or hyper-thyroidism
* Have an initiation, a cessation or change of dose (up to three weeks prior to the study's start) of any chronic medications or dietary supplements or any planned change of chronic medications or dietary supplements during the study;
* Have implanted (e.g., surgical clips or staples) metal objects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female breast cancer survivors
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Compare peripheral immune markers (cytokines), C-reactive protein levels and brain neurotransmitters (glutamate, GABA, myoinositol, and resting state intrinsic connectivity). | 6 weeks

SECONDARY OUTCOMES:
Compare fatigue, pain, and sleep quality with peripheral immune markers, CRP, and brain markers. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States